CLINICAL TRIAL: NCT04359199
Title: QUantitative Assessment of Swallowing After Radiation (QUASAR): A Longitudinal Comparison of Swallowing Function by Systemic Therapy in Head and Neck Cancer Patients
Brief Title: QUantitative Assessment of Swallowing After Radiation (QUASAR)
Acronym: QUASAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Loren Mell, MD (Other)
Responsible Party: Sponsor-Investigator, Loren Mell, MD, Director, Division of Clinical and Translational Research/ Department of Radiation Medicine and Applied Sciences, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 190048
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer; Dysphagia; Oropharyngeal Dysphagia; Oropharynx Cancer; Oropharynx Squamous Cell Carcinoma
Keywords: head and neck cancer; oropharyngeal dysphagia; radiation therapy; immunotherapy; videofluoroscopic swallow study; modified barium swallow study; oropharynx cancer; oropharynx squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Cetuximab; Drug Therapy; Cisplatin; Immunotherapy; pembrolizumab; Nivolumab; durvalumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiotherapy with chemotherapy: Patients treated with definitive RT and chemotherapy (cisplatin) or targeted therapy (cetuximab)
  Interventions: Radiation: Radiation Therapy; Drug: Cetuximab; Drug: Chemotherapy
- Radiotherapy with immunotherapy: Patients treated with definitive RT and immunotherapy (pembrolizumab, nivolumab, or durvalumab)
  Interventions: Radiation: Radiation Therapy; Drug: Immunotherapy

INTERVENTIONS:
Radiation: Radiation Therapy — Routine radiation dosing (approximately 70 Gy in 35 fractions over 6.5 weeks) to the head and neck for the treatment of head and neck cancer
  Other Names: radiotherapy; RT
Drug: Cetuximab — Cetuximab is an epidermal growth factor receptor (EGFR) inhibitor used for the treatment of head and neck cancer
  Other Names: Erbitux
  Groups: Radiotherapy with chemotherapy
Drug: Chemotherapy — Cisplatin is a chemotherapy medication used to treat a number of cancers, including head and neck cancer
  Other Names: Cisplatin
  Groups: Radiotherapy with chemotherapy
Drug: Immunotherapy — Keytruda or Pembrolizumab is a highly selective humanized monoclonal IgG4 antibody directed against the PD-1 receptor on the cell surface.
  Opdivo or Nivolumab is a targeted therapy. It is a human programmed death receptor-1 (PD-1) blocking antibody.
  Imfinzi or Durvalumab is an anti-cancer ("antineoplastic") drug. This medication is classified as an Anti-PD-L1 monoclonal antibody.
  Other Names: pembrolizumab; Keytruda; nivolumab; Opdivo; durvalumab; Imfinzi
  Groups: Radiotherapy with immunotherapy

SUMMARY:
To use novel methods for quantitative analysis of VFSS (videofluoroscopic swallow study, also known as modified barium swallow) to study and compare dysphagia in patients treated for head and neck carcinoma with concurrent radiation therapy and chemotherapy (cisplatin) or targeted therapy (cetuximab) vs. immunotherapy (pembrolizumab, nivolumab, or durvalumab).

Our hypothesis is that pharyngeal constriction will be greater (lower ratio) with concurrent immunotherapy compared to chemotherapy, as measured by the pharyngeal constriction ratio (PCR).

DETAILED DESCRIPTION:
The QUASAR study will use a prospective, observational, cross sectional design (See Schema). HNC patients treated with definitive RT and immunotherapy or chemotherapy (cetuximab or cisplatin) will undergo VFSS at 4-6 and 12-24 months post-treatment. Patients enrolled prior to 6 months after finishing therapy will undergo a swallow study during the 4-6 month period AND the 12-24 month period. Patients enrolled after 6 months after finishing therapy will undergo a single swallow study in the 12-24 month period. The primary endpoint of PCR at 12-24 months will be compared between patients treated with immunotherapy versus chemotherapy.

All patients with HNC treated with definitive RT and systemic therapy at our institution will be eligible. In particular, we will recruit patients for this study from participants in two ongoing trials investigating the use of concurrent immunotherapy. The KEYCHAIN trial (ClinicalTrials.gov Identifier: NCT03383094) randomizes patients with locally advanced p16+ HNC undergoing definitive RT to concurrent q3 week cisplatin versus concurrent and adjuvant pembrolizumab. NRG-HN004 (ClinicalTrials.gov Identifier: NCT03258554) is a cooperative group trial that compares HNC patients that are not eligible for cisplatin undergoing definitive radiation therapy to concurrent cetuximab versus durvalumab.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven, un-resected invasive carcinoma of the head and neck.
* Treated with definitive RT and concurrent systemic therapy or treated within the past 4-24 months
* Concurrent systemic therapy with Cisplatin, Cetuximab or immunotherapy.
* Age ≥ 18
* Able to understand and willing to sign a written informed consent.

Exclusion Criteria:

* Prior radiotherapy that would result in overlap of planned radiation therapy fields.
* Prior systemic chemotherapy, unless as part of the coordinated plan of care for the treatment of the carcinoma (e.g., induction/neoadjuvant chemotherapy is allowed)
* Planned adjuvant (i.e., following definitive chemoradiotherapy) chemotherapy or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck carcinoma treated with definitive radiation therapy and systemic therapy (chemotherapy or immunotherapy) in the University of California San Diego Healthcare System will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Swallowing function 12-24 months after concurrent radiation and systemic therapy for HNC, as measured by the PCR | 12-24 months
  will use a two-sample t-test at 0.05 level to compare Pharyngeal Constriction Ratio (PCR) between groups

SECONDARY OUTCOMES:
Quantitative swallowing function at 4-6 months and 12-24 months by PCR, TPT, PRR and PPWT | 4-6 months and 12-24 months
  To compare swallowing function between systemic therapies with additional quantitative metrics of swallowing dysfunction from the VFSS including TPT, PRR and PPWT.
  The presence of aspiration or strictures on VFSS will be compared as binary variables between groups using Pearson's Chi squared test.
Correlation between quantitative swallowing function and patient reported symptoms using the EAT-10 tool | 12-24 months
  To compare patient reported assessments of swallowing function with the EAT-10 tool between systemic therapies.
  To test if there is correlation between the quantitative VFSS metrics and patient reported outcomes on the EAT-10 index, we will calculate Pearson's correlation coefficient and plot the results on a correlation matrix. The Holm step down procedure will be used to adjust for multiple testing to control the family-wise error rate at 0.05 level.
Correlation between radiation dose and location of swallowing function and quantitative swallowing function | 24 months
  The purpose of this aim is to evaluate the effect of radiation dose on swallowing structures, applying a previously developed space-preserving NTCP approach based on principal component analysis (PCA).
  Using this approach, dose distributions to the global swallowing apparatus (i.e. pharynx, larynx and esophagus) will be standardized for patients from both arms of Aim 1, using deformable registration to standardize organs and 3-D dose distributions to a common template. Dose distributions will be converted into a dose array and PCA will be applied to the dose array, as previously described. We will then use PC linear regression to identify eigenvectors significantly associated with long term dysphagia (as measured by PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Loren K Mell, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCSD Moores Cancer Center, La Jolla, California

REFERENCES:
- [Background] Naidoo J, Page DB, Li BT, Connell LC, Schindler K, Lacouture ME, Postow MA, Wolchok JD. Toxicities of the anti-PD-1 and anti-PD-L1 immune checkpoint antibodies. Ann Oncol. 2015 Dec;26(12):2375-91. doi: 10.1093/annonc/mdv383. Epub 2015 Sep 14. PMID 26371282
- [Background] Basch E, Iasonos A, McDonough T, Barz A, Culkin A, Kris MG, Scher HI, Schrag D. Patient versus clinician symptom reporting using the National Cancer Institute Common Terminology Criteria for Adverse Events: results of a questionnaire-based study. Lancet Oncol. 2006 Nov;7(11):903-9. doi: 10.1016/S1470-2045(06)70910-X. PMID 17081915
- [Background] Leonard R, Kendall K. Dysphagia Assessment and Treatment Planning: A Team Approach. Fourth. Plural Publishing; 2018
- [Background] Stoeckli SJ, Huisman TA, Seifert B, Martin-Harris BJ. Interrater reliability of videofluoroscopic swallow evaluation. Dysphagia. 2003 Winter;18(1):53-7. doi: 10.1007/s00455-002-0085-0. PMID 12497197
- [Background] Yip H, Leonard R, Belafsky PC. Can a fluoroscopic estimation of pharyngeal constriction predict aspiration? Otolaryngol Head Neck Surg. 2006 Aug;135(2):215-7. doi: 10.1016/j.otohns.2006.03.016. PMID 16890070
- [Background] Leonard R, Rees CJ, Belafsky P, Allen J. Fluoroscopic surrogate for pharyngeal strength: the pharyngeal constriction ratio (PCR). Dysphagia. 2011 Mar;26(1):13-7. doi: 10.1007/s00455-009-9258-4. Epub 2009 Oct 24. PMID 19856026
- [Background] Servagi-Vernat S, Ali D, Roubieu C, Durdux C, Laccourreye O, Giraud P. Dysphagia after radiotherapy: state of the art and prevention. Eur Ann Otorhinolaryngol Head Neck Dis. 2015 Feb;132(1):25-9. doi: 10.1016/j.anorl.2013.09.006. Epub 2014 Jun 9. PMID 24924114
- [Background] Jensen K, Lambertsen K, Grau C. Late swallowing dysfunction and dysphagia after radiotherapy for pharynx cancer: frequency, intensity and correlation with dose and volume parameters. Radiother Oncol. 2007 Oct;85(1):74-82. doi: 10.1016/j.radonc.2007.06.004. Epub 2007 Jul 27. PMID 17673322
- [Background] Duprez F, Madani I, De Potter B, Boterberg T, De Neve W. Systematic review of dose--volume correlates for structures related to late swallowing disturbances after radiotherapy for head and neck cancer. Dysphagia. 2013 Sep;28(3):337-49. doi: 10.1007/s00455-013-9452-2. Epub 2013 Feb 22. PMID 23429941
- [Background] Liang Y, Messer K, Rose BS, Lewis JH, Jiang SB, Yashar CM, Mundt AJ, Mell LK. Impact of bone marrow radiation dose on acute hematologic toxicity in cervical cancer: principal component analysis on high dimensional data. Int J Radiat Oncol Biol Phys. 2010 Nov 1;78(3):912-9. doi: 10.1016/j.ijrobp.2009.11.062. Epub 2010 May 14. PMID 20472344
- [Result] Green G, Kim E, Carmona R, Shen H, Murphy JD, Mell LK. Incidence of Long-Term Esophageal Dilation With Various Treatment Approaches in the Older Head and Neck Cancer Population. Front Oncol. 2018 Oct 23;8:466. doi: 10.3389/fonc.2018.00466. eCollection 2018. PMID 30406032